CLINICAL TRIAL: NCT03222973
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study With Optional Open-Label Extension in Subjects With Relapsing Multiple Sclerosis to Evaluate the Efficacy and Safety of BIIB033 as an Add-On Therapy to Anti-Inflammatory Disease-Modifying Therapies
Brief Title: Efficacy and Safety of BIIB033 (Opicinumab) as an Add-on Therapy to Disease-Modifying Therapies (DMTs) in Relapsing Multiple Sclerosis (MS)
Acronym: AFFINITY
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The top-line results from the Part 1 did not meet the pre-specified primary endpoint nor the key secondary endpoints. The decision to discontinue study 215MS202 Part 2 was not based on safety concerns.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 215MS202; 2017-001224-22 (EudraCT Number)
Record Dates: First submitted 2017-07-17; First posted 2017-07-19 (Actual); Results first posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-03

CONDITIONS: Multiple Sclerosis
Keywords: Remyelination; Re-myelination; DMT; LINGO-1; Anti-LINGO-1; Opicinumab
MeSH Terms: conditions — Multiple Sclerosis | interventions — opicinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BIIB033 (opicinumab) 750 mg (Experimental): Participants with relapsing multiple sclerosis (RMS) will receive BIIB033 750 milligram (mg) intravenously (IV) as an add-on therapy to a background disease-modifying therapy (DMT) once every 4 weeks over 72 weeks in Part 1 and once every 4 weeks over 96 weeks in Part 2.
  Interventions: Drug: BIIB033 (opicinumab)
- Placebo (Placebo Comparator): Participants with RMS will receive placebo IV as an add-on therapy to a background DMT once every 4 weeks over 72 weeks in Part 1 and BIIB033 once every 4 weeks over 96 weeks in Part 2. The placebo looks like BIIB033 but does not contain the active ingredient that is thought to have an effect on MS disease. The placebo used in this study is sterile normal saline (water with a small amount of sodium chloride [salt]).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIB033 (opicinumab) — Administered as specified in the treatment arm
  Arms: BIIB033 (opicinumab) 750 mg
Drug: Placebo — Administered as specified in the treatment arm
  Arms: Placebo

SUMMARY:
The primary objective of Part 1 of this study is to evaluate the effects of BIIB033 versus placebo on disability improvement over 72 weeks. The primary objective of Part 2 of this study is to evaluate the long-term safety profile of BIIB033 as an add-on therapy in participants with MS.

The secondary objective of Part 1 is to evaluate the effects of BIIB033 versus placebo on additional measures of disability improvement. The secondary objective of Part 2 is to investigate long-term efficacy (disability improvement) and additional safety measures of BIIB033 as an add-on therapy in participants with MS.

ELIGIBILITY:
Key Inclusion Criteria: Part 1

* Baseline Expanded Disability Status Scale (EDSS) of 2.0 to 6.0, have a diagnosis of relapsing-remitting multiple sclerosis (RRMS) per the 2010 McDonald's criteria or onset of secondary progressive multiple sclerosis (SPMS) per the Lublin and Reingold criteria, and should have experienced their first MS symptom(s) within the previous 20 years.
* Subjects must have experienced at least 1 of the following within 24 months prior to Day 1/Baseline: a clinical relapse (but not within 24 weeks prior to Day 1/Baseline), gadolinium-enhancing lesions on brain or spinal cord magnetic resonance imaging (MRI), or new T2 lesion(s) on brain or spinal cord MRI.
* Subjects must be on a stable dose of a protocol-specified anti-inflammatory disease-modifying therapy (DMT) (IFNβ [Avonex, Plegridy, Betaferon/Betaseron, or Rebif], dimethyl fumarate (DMF) [Tecfidera], or natalizumab [Tysabri]) for at least 24 weeks prior to enrollment.
* In addition, subjects must have met protocol-defined MRI characteristics using magnetization transfer ratio (MTR) and diffusion tensor imaging (DTI) sequences at Screening/Baseline.

Key Inclusion Criteria: Part 2

-Subjects who complete study treatment (BIIB033 or placebo) at Part 1/Week 72 Visit.

Key Exclusion Criteria: Part 1

* Primary progressive MS
* An MS relapse that has occurred within 24 weeks prior to Day 1/Baseline or the subject has not stabilized from a previous relapse at the time of Screening.
* Treatment with any chemotherapeutic agents (e.g., mitoxantrone, cyclophosphamide, cladribine), cell-depleting monoclonal antibodies (mAbs) (e.g., rituximab, ocrelizumab, alemtuzumab), total lymphoid irradiation, T-cell or T-cell receptor vaccination, or teriflunomide within 1 year prior to Day 1/Baseline.
* Treatment with other anti-inflammatory DMTs (e.g., GA, fingolimod, daclizumab) or plasmapheresis within 24 weeks prior to Day1/Baseline.
* Treatment with Botox for limb spasticity within 24 weeks before Day 1/Baseline.
* Contraindications to MRI, for example, presence of pacemakers or other implanted metal devices (excluding dental braces), an allergy to gadolinium renal impairment, or claustrophobia that cannot be medically managed.
* History of human immunodeficiency virus or other immunodeficient conditions.
* History of malignancy; however, subjects with a history of excised or treated basal cell carcinoma or fewer than 3 squamous cell carcinomas are eligible to participate in this study.

Key Exclusion Criteria: Part 2

* Subjects who did not complete study treatment in Part 1/Week 72 Visit
* Subjects who have a duration >12 weeks between their Part 1/Week 72 Visit and Part 2/Day 1.
* Contraindications to MRI, for example, presence of pacemakers or other implanted metal devices (excluding dental braces), an allergy to Gd, renal impairment, or claustrophobia that cannot be medically managed.
* History of human immunodeficiency virus or other immunodeficient conditions not related to DMT treatment.
* History of malignancy unless enrollment is approved by the Sponsor; subjects with a history of excised or treated basal cell carcinoma or fewer than 3 squamous cell carcinomas are eligible to participate in this study.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 263 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2021-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (144):
- United States (47):
  - Research Site, Cullman, Alabama
  - Research Site, Gilbert, Arizona
  - Research Site, Berkeley, California
  - Research Site, Long Beach, California
  - Research Site, Newport Beach, California
  - Research Site, Orange, California
  - Research Site, Centennial, Colorado
  - Research Site, Fort Collins, Colorado
  - Research Site, Stamford, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Sunrise, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Overland Park, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Lexington, Massachusetts
  - Research Site, Wellesley, Massachusetts
  - Research Site, Farmington Hills, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Freehold, New Jersey
  - Research Site, Teaneck, New Jersey
  - Research Site, Latham, New York
  - Research Site, New York, New York
  - Research Site, Patchogue, New York
  - Research Site, Rochester, New York
  - Research Site, Stony Brook, New York
  - Research Site, Durham, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Willow Grove, Pennsylvania
  - Research Site, Knoxville, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Round Rock, Texas
  - Research Site, Orem, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Seattle, Washington
- Australia (7):
  - Research Site, Box Hill, Victoria
  - Research Site, Clayton, Victoria
  - Research Site, Heidelberg, Victoria
  - Research Site, Melbourne, Victoria
  - Research Site, Parkville, Victoria
  - Research Site, New Lambton Heights
  - Research Site, Westmead
- Belgium (6):
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, La Louvière
  - Research Site, Leuven
  - Research Site, Roeselare
- Canada (8):
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Gatineau, Quebec
  - Research Site, Longueuil, Quebec
  - Research Site, Montreal, Quebec
- Czechia (5):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Jihlava
  - Research Site, Pardubice
  - Research Site, Prague
- France (11):
  - Research Site, Strasbourg, Bas Rhin
  - Research Site, Nîmes, Gard
  - Research Site, Bordeaux, Gironde
  - Research Site, Toulouse, Haute Garonne
  - Research Site, Montpellier, Herault
  - Research Site, Nantes, Loire Atlantique
  - Research Site, Lille, Nord
  - Research Site, Clermont-Ferrand, Puy De Dome
  - Research Site, Bron, Rhone
  - Research Site, Amiens, Somme
  - Research Site, Paris
- Germany (10):
  - Research Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Research Site, Tübingen, Baden-Wurttemberg
  - Research Site, Ulm, Baden-Wurttemberg
  - Research Site, Munich, Bavaria
  - Research Site, Bochum, North Rhine-Westphalia
  - Research Site, Düsseldorf, North Rhine-Westphalia
  - Research Site, Trier, Rhineland-Palatinate
  - Research Site, Dresden, Saxony
  - Research Site, Berlin
  - Research Site, Münster
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Esztergom
  - Research Site, Kistarcsa
  - Research Site, Pécs
- Research Site, Ramat Gan, Israel
- Italy (10):
  - Research Site, Montichiari, Brescia
  - Research Site, Pozzilli, Isernia
  - Research Site, Cefalù, Palermo
  - Research Site, Genova
  - Research Site, Messina
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Verona
- Research Site, Geleen, Netherlands
- Poland (9):
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Szczecin
  - Research Site, Warsaw
  - Research Site, Zabrze
- Spain (7):
  - Research Site, Salt, Girona
  - Research Site, Majadahonda, Madrid
  - Research Site, Barakaldo, Vizcaya
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Madrid
  - Research Site, Seville
- Switzerland (5):
  - Research Site, Aarau
  - Research Site, Basel
  - Research Site, Bern
  - Research Site, Lugano
  - Research Site, Zurich
- United Kingdom (13):
  - Research Site, Exeter, Devon
  - Research Site, Plymouth, Devon
  - Research Site, London, Greater London
  - Research Site, Salford, Greater Manchester
  - Research Site, Liverpool, Merseyside
  - Research Site, Nottingham, Nottinghamshire
  - Research Site, Oxford, Oxfordshire
  - Research Site, Glasgow, Strathclyde
  - Research Site, Newcastle upon Tyne, Tyne & Wear
  - Research Site, Leeds, West Yorkshire
  - Research Site, Brighton
  - Research Site, Sheffield
  - Research Site, Swansea

REFERENCES:
- [Derived] Calabresi PA, Giovannoni G, Hartung HP, Naismith RT, Fox RJ, Sormani MP, Arnold DL, Kappos L, Valis M, Newsome SD, Belkin MI, Bartholome E, Riester K, Javor A, Lyons J, Bradley DP, Fisher E, Tagge I, Naylor ML, Belachew S, Deykin A, Franchimont N, Zhu B, Cheng W. Safety and efficacy of opicinumab in participants with relapsing multiple sclerosis (AFFINITY Part 1): A randomized, controlled, phase 2 trial. Mult Scler. 2026 Jan;32(1):107-120. doi: 10.1177/13524585251396433. Epub 2025 Dec 26. PMID 41454463
- [Derived] Elliott C, Rudko DA, Arnold DL, Fetco D, Elkady AM, Araujo D, Zhu B, Gafson A, Tian Z, Belachew S, Bradley DP, Fisher E. Lesion-level correspondence and longitudinal properties of paramagnetic rim and slowly expanding lesions in multiple sclerosis. Mult Scler. 2023 May;29(6):680-690. doi: 10.1177/13524585231162262. Epub 2023 Apr 10. PMID 37036134
- [Derived] Hanf KJM, Arndt JW, Liu Y, Gong BJ, Rushe M, Sopko R, Massol R, Smith B, Gao Y, Dalkilic-Liddle I, Lee X, Mojta S, Shao Z, Mi S, Pepinsky RB. Functional activity of anti-LINGO-1 antibody opicinumab requires target engagement at a secondary binding site. MAbs. 2020 Jan-Dec;12(1):1713648. doi: 10.1080/19420862.2020.1713648. PMID 31928294

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at the investigative sites in the Australia, Belgium, Canada, Czech Republic, France, Germany, Hungary, Israel, Italy, Netherlands, Poland, Spain, Switzerland, United Kingdom and United States from 15 November 2017 to 12 February 2021.
Pre-assignment Details: A total of 263 participants with relapsing multiple sclerosis (RMS) were randomized in Part 1 (Placebo-controlled) of the study to receive BIIB033 or placebo. Participants who completed Part 1 and were eligible were enrolled into Part 2 (Open-label) of the study to receive BIIB033. Part 2 of the study was terminated early based on Sponsor's decision.
Groups:
- Part 1: Placebo: Participants with RMS received placebo intravenously (IV) as an add-on therapy to a background disease-modifying therapy (DMT) once every 4 weeks over 72 weeks.
- Part 1: BIIB033 750 mg: Participants with RMS received BIIB033 750 milligrams (mg) IV as an add-on therapy to a background DMT once every 4 weeks over 72 weeks.
- Part 2: Placebo to BIIB033 750 mg: Participants who received placebo and completed Part 1 were enrolled into Part 2 to receive BIIB033 750 mg IV as an add-on therapy to a background DMT once every 4 weeks for up to a maximum of 80 weeks.
- Part 2: BIIB033 750 mg: Participants who received BIIB033 and completed Part 1 were enrolled into Part 2 to receive BIIB033 750 mg IV as an add-on therapy to a background DMT once every 4 weeks for up to a maximum of 77 weeks.
Period: Part 1 (Week 0 to Week 72)
Arm/Group | Part 1: Placebo | Part 1: BIIB033 750 mg | Part 2: Placebo to BIIB033 750 mg | Part 2: BIIB033 750 mg
Started | 131 | 132 | 0 | 0
Intent-to-treat (ITT) Population | 131 | 132 | 0 | 0
Safety Population | 131 | 132 | 0 | 0
Completed | 107 | 118 | 0 | 0
Not Completed | 24 | 14 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0
Not completed — Consent Withdrawn | 12 | 9 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0
Not completed — Other | 8 | 2 | 0 | 0
Period: Part 2 (Week 73 to Week 168)
Arm/Group | Part 1: Placebo | Part 1: BIIB033 750 mg | Part 2: Placebo to BIIB033 750 mg | Part 2: BIIB033 750 mg
Started | 0 | 0 | 101 (6 participants who completed Part 1 did not enter Part 2.) | 113 (5 participants who completed Part 1 did not enter Part 2.)
ITT Population | 0 | 0 | 100 | 113
Safety Population | 0 | 0 | 100 | 113
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 101 | 113
Not completed — Adverse Event | 0 | 0 | 2 | 0
Not completed — Consent Withdrawn | 0 | 0 | 10 | 11
Not completed — Investigator Decision | 0 | 0 | 2 | 1
Not completed — Pregnancy | 0 | 0 | 2 | 1
Not completed — Other | 0 | 0 | 84 | 100
Not completed — Participants Not Dosed | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants who received at least 1 dose of study treatment. Participants were analyzed according to their treatment assignment regardless of actual treatment received.
Groups:
- Part 1: Placebo: Participants with RMS received placebo IV as an add-on therapy to a background DMT once every 4 weeks over 72 weeks.
- Part 1: BIIB033 750 mg: Participants with RMS received BIIB033 750 mg IV as an add-on therapy to a background DMT once every 4 weeks over 72 weeks.
- Total: Total of all reporting groups
Arm/Group | Part 1: Placebo | Part 1: BIIB033 750 mg | Total
Number analyzed (Participants) | 131 | 132 | 263
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (9.25) | 39.4 (9.12) | 38.6 (9.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 90 | 169
  Male | 52 | 42 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 13 | 18
  Not Hispanic or Latino | 123 | 116 | 239
  Unknown or Not Reported | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 10 | 14
  White | 122 | 118 | 240
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Overall Response Score
Description: Overall Response Score is a multicomponent score based on 4 components: Expanded Disability Status Scale (EDSS), Timed 25-Foot Walk (T25FW), 9-Hole Peg Test in the dominant hand (9HPT-D), and 9HPT in the nondominant hand (9HPT-ND). Overall Score was sum of 4 components at each visit and ranges from +4 (improvement) to -4 (worsening). At each visit, each component is given a score relative to baseline (BL): -1 if threshold is met for worsening, 0 if no changes meet threshold criteria, or +1 if threshold is met for improvement. For T25FW and 9HPT improvement is ≥15% decrease in time from BL and worsening is ≥15% increase in time from BL. For EDSS, improvement is: ≥1.0-point decrease in EDSS from a BL score of ≤6.0, and worsening is defined as a ≥1-point increase from a BL score of ≤5.5 or a ≥0.5-point increase from a BL score equal to 6.0. Positive Overall Response Score indicated that there was improvement in more components than there was worsening.
Time Frame: Part 1: Baseline to Week 72
Population: ITT population included all randomized participants who received at least 1 dose of study treatment. Participants were analyzed according to their treatment assignment regardless of actual treatment received.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Part 1: Placebo | Part 1: BIIB033 750 mg
Number analyzed (Participants) | 131 | 132
score on a scale | -0.04 [-0.18 to 0.11] | 0.11 [-0.03 to 0.25]
Statistical Analysis 1: Comparison: Part 1: Placebo vs Part 1: BIIB033 750 mg; Over 72 weeks: Overall Response Score; Test type: Superiority; p = 0.1479, MMRM — P-values are based on the Mixed Model for Repeated Measures (MMRM) adjusted for background DMT group, baseline magnetization transfer ratio (MTR)/diffusion tensor imaging (DTI) category and baseline component assessments; Treatment Difference = 0.15, 95% CI 2-sided [-0.05 to 0.35]

2. Primary Outcome: Part 2: Number of Participants Experiencing Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A SAE is any untoward medical occurrence that at any dose results in death, life-threatening event, requires inpatient hospitalization, significant disability/incapacity or congenital anomaly.
Time Frame: Part 2: Baseline to Week 169
Population: Safety population included all participants who received at least 1 dose of study treatment. Participants were analyzed based on the actual treatment allocation.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo to BIIB033 750 mg | Part 2: BIIB033 750 mg
Number analyzed (Participants) | 100 | 113
Participants
  AEs | 71 | 76
  SAEs | 9 | 2

3. Secondary Outcome: Part 1: Percentage of Participants With 12-week Confirmed Improvement in at Least 1 of the Following Assessments: EDSS, T25FW, 9HPT-D, or 9HPT-ND
Description: EDSS measures disability status over time in MS on a scale ranging from 0 to 10, with higher scores indicating more disability. For EDSS, improvement is defined as a ≥1.0-point decrease in EDSS from a BL score of ≤6.0. T25FW is a quantitative mobility and leg function performance test based on a timed walk over 25 feet that is averaged between two completed trials. Longer time indicates slower walking. The 9HPT is a quantitative test of upper extremity function that measures the time it takes to place 9 pegs into 9 holes and then remove the pegs. Longer time indicates poorer upper limb function. For T25FW and 9HPT ≥15% decrease in time from BL indicates improvement.
Time Frame: Part 1: Baseline to Week 72
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Placebo | Part 1: BIIB033 750 mg
Number analyzed (Participants) | 131 | 132
percentage of participants | 37 | 39
Statistical Analysis 1: Comparison: Part 1: Placebo vs Part 1: BIIB033 750 mg; Test type: Superiority; p = 0.7682, Regression, Logistic — Odds ratio (active vs. placebo), 95% CI and p-value are based on logistic regression adjusted for background DMT group, baseline MTR/DTI category and baseline component assessments; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.65 to 1.79]

4. Secondary Outcome: Part 1: Percentage of Participants With 12-week Confirmed Improvement in at Least 1 of the Following Assessments: EDSS, T25FW, 9HPT-D, 9HPT-ND, or 3-Second Paced Auditory Serial Addition Test (PASAT-3)
Description: EDSS measures disability status over time in MS (scale range: 0-10), higher scores=more disability and improvement defined as ≥1.0-point decrease in EDSS from BL score ≤6.0. T25FW is quantitative mobility and leg function performance test, where timed walk over 25 feet that is averaged between two completed trials. Longer time=slower walking. 9HPT is quantitative test of upper extremity function, measures time to place 9 pegs into 9 holes and then remove pegs. Longer time=poorer upper limb function. PASAT assesses auditory information processing speed. In 3-second PASAT, numbers are presented at a rate of 1 every 3 seconds with scores (range 0-120), higher scores=better working memory. For T25FW and 9HPT ≥15% decrease in time from BL is improvement. For PASAT ≥15% increase from BL is improvement.
Time Frame: Part 1: Baseline to Week 72
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Placebo | Part 1: BIIB033 750 mg
Number analyzed (Participants) | 131 | 132
percentage of participants | 60 | 52
Statistical Analysis 1: Comparison: Part 1: Placebo vs Part 1: BIIB033 750 mg; Test type: Superiority; p = 0.2131, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.41 to 1.22]

5. Secondary Outcome: Part 1: Percentage of Participants With 12-week Confirmed Improvement in at Least 1 of the Following Assessments: EDSS, T25FW, 9HPT-D, or 9HPT-ND, and Without Confirmed Worsening in Any of the 4 Assessments During the 72 Weeks of the Study
Description: EDSS measures disability status over time in MS on a scale ranging from 0 to 10, with higher scores indicating more disability. For EDSS, improvement is defined as a ≥1.0-point decrease in EDSS from a BL score of ≤6.0, and worsening is defined as a ≥1-point increase from a BL score of ≤5.5 or a ≥0.5-point increase from a BL score equal to 6.0. T25FW is a quantitative mobility and leg function performance test based on a timed walk over 25 feet that is averaged between two completed trials. Longer time indicates slower walking. The 9HPT is a quantitative test of upper extremity function that measures the time it takes to place 9 pegs into 9 holes and then remove the pegs. Longer time indicates poorer upper limb function. For T25FW and 9HPT ≥15% decrease in time from BL indicates improvement and ≥15% increase in time from BL indicates worsening.
Time Frame: Part 1: Baseline to Week 72
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Placebo | Part 1: BIIB033 750 mg
Number analyzed (Participants) | 131 | 132
percentage of participants | 31 | 28
Statistical Analysis 1: Comparison: Part 1: Placebo vs Part 1: BIIB033 750 mg; Test type: Superiority; p = 0.4654, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.47 to 1.41]

6. Secondary Outcome: Part 1: Percentage of Participants With 12-week Confirmed Improvement in at Least 1 of the Following Assessments: EDSS, T25FW, 9HPT-D, 9HPT-ND, and Symbol Digit Modalities Test (SDMT)
Description: EDSS measures disability status over time in MS on a scale (range 0-10), higher scores=more disability. For EDSS, improvement is: a ≥1.0-point decrease in EDSS from a BL score of ≤6.0. T25FW is a quantitative mobility and leg function performance test based on a timed walk over 25 feet that is averaged between two completed trials. Longer time=slower walking. 9HPT is quantitative test of upper extremity function that measures time it takes to place 9 pegs into 9 holes and then remove pegs. Longer time=poorer upper limb function. For T25FW and 9HPT ≥15% decrease in time from BL indicates improvement. The SDMT measures time to pair abstract geometric symbols with specific numbers. The score is the number of correctly coded items (range 0-110) in 90 seconds, higher scores=better outcome. Improvement is: ≥4-point increase from BL.
Time Frame: Part 1: Baseline to Week 72
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Placebo | Part 1: BIIB033 750 mg
Number analyzed (Participants) | 131 | 132
percentage of participants | 63 | 75
Statistical Analysis 1: Comparison: Part 1: Placebo vs Part 1: BIIB033 750 mg; Test type: Superiority; p = 0.0417, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.78, 95% CI 2-sided [1.02 to 3.11]

7. Secondary Outcome: Part 1: Percentage of Participants With 12-week Confirmed Improvement in at Least 1 of the Following Assessments: EDSS, T25FW, 9HPT-D, or 9HPT-ND (20% Thresholds for T25FW and 9HPT)
Description: as for outcome 3
Time Frame: Part 1: Baseline to Week 72
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Placebo | Part 1: BIIB033 750 mg
Number analyzed (Participants) | 131 | 132
percentage of participants | 25 | 32
Statistical Analysis 1: Comparison: Part 1: Placebo vs Part 1: BIIB033 750 mg; Test type: Superiority; p = 0.2908, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.78 to 2.33]

8. Secondary Outcome: Part 2: Overall Response Score
Time Frame: Part 2: Baseline to Week 96
Population: Part 1 of Study 215MS202 failed to meet its primary endpoint of ORS over 72 weeks. Trial also failed to show efficacy in its secondary endpoints. Thus, Sponsor decided to terminate Part 2 of study early, and no participants had the opportunity to complete Part 2 of the study. No data was collected as per the protocol prespecified Part 2 efficacy analyses to assess the long-term efficacy of BIIB033 in Part 2.
Arm/Group | Part 2: Placebo to BIIB033 750 mg | Part 2: BIIB033 750 mg
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Part 2: Percentage of Participants With 24-week Confirmed Improvement in at Least 1 of the Following Assessments: EDSS, T25FW, 9HPT-D, or 9HPT-ND
Time Frame: Part 2: Baseline to Week 108
Population: as for outcome 8
Arm/Group | Part 2: Placebo to BIIB033 750 mg | Part 2: BIIB033 750 mg
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Part 2: Percentage of Participants With 24-week Confirmed Improvement in at Least 1 of the Following Assessments: EDSS, T25FW, 9HPT-D, 9HPT-ND, or PASAT-3
Time Frame: Part 2: Baseline to Week 108
Population: as for outcome 8
Arm/Group | Part 2: Placebo to BIIB033 750 mg | Part 2: BIIB033 750 mg
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Part 2: Percentage of Participants With 24-week Confirmed Improvement in at Least 1 of the Following Assessments: EDSS, T25FW, 9HPT-D, or 9HPT-ND, and Without Confirmed Worsening in Any of the 4 Assessments During the 96 Weeks of the Study
Time Frame: Part 2: Baseline to Week 96
Population: as for outcome 8
Arm/Group | Part 2: Placebo to BIIB033 750 mg | Part 2: BIIB033 750 mg
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Part 2: Percentage of Participants With 24-week Confirmed Improvement in at Least 1 of the Following Assessments: EDSS, T25FW, 9HPT-D, 9HPT-ND, and SDMT
Time Frame: Part 2: Baseline to Week 108
Population: as for outcome 8
Arm/Group | Part 2: Placebo to BIIB033 750 mg | Part 2: BIIB033 750 mg
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Part 2: Percentage of Participants With 24-week Confirmed Improvement in at Least 1 of the Following Assessments: EDSS, T25FW, 9HPT-D, or 9HPT-ND (20% Thresholds for T25FW and 9HPT)
Time Frame: Part 2: Baseline to Week 108
Population: as for outcome 8
Arm/Group | Part 2: Placebo to BIIB033 750 mg | Part 2: BIIB033 750 mg
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Part 2: Number of Participants With Potentially Clinically Significant Abnormal Laboratory Values
Description: Laboratory assessments including hematology and blood chemistry were evaluated for safety. Criteria for abnormality: In 10^9/liter (L) [white blood cells <3.0/>16, neutrophils <1.5/ >13.5, lymphocytes <0.8/ >12, monocytes >2.5, eosinophils >1.6, basophils >1.6, platelets <=75/ >=700], hemoglobin <=95 [female (F)] or <=115 [male (M)] or >=175 (F) or >=190 (M) gram per liter (g/L), hematocrit <=32 (F) or <=37 (M) or >=54 (F) or >=60 (M) percentage (%), red blood cells <=3.5/ >=6.4 10^12/L, in millimoles per liter (mmol/L) [sodium <=126/ >=156, potassium <=3/ >=6, chloride <=90/ >=118, bicarbonate <=16/ >=35, calcium <=2/ >=3, phosphorous <=0.5491/ >=1.7119, glucose (non-fasting) <=2.2/>=13.75], AST/SGOT >=3x upper limit of normal (ULN), ALT/SGPT >=3xULN, alkaline phosphatase >=3xULN, creatinine >=1.5xULN, total bilirubin >=1.5xULN, total protein <=45/ >=100 g/L, albumin <=25 g/L, uric acid >=501.5 (F)/>=619.5 (M) micromole (umol)/L
Time Frame: Part 2: Baseline to Week 96
Population: Safety population included all participants who received at least 1 dose of study treatment. Participants were analyzed based on the actual treatment allocation. 'Number Analyzed' signifies number of participants analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo to BIIB033 750 mg | Part 2: BIIB033 750 mg
Number analyzed (Participants) | 100 | 113
Participants
  White blood cells [10^9/L]: <3.0: number analyzed (Participants) | 98 | 113
  White blood cells [10^9/L]: <3.0 | 3 | 3
  White blood cells (10^9/L): >16: number analyzed (Participants) | 98 | 113
  White blood cells (10^9/L): >16 | 2 | 0
  Neutrophils (10^9/L): <1.5: number analyzed (Participants) | 98 | 113
  Neutrophils (10^9/L): <1.5 | 3 | 3
  Neutrophils (10^9/L): >13.5: number analyzed (Participants) | 98 | 113
  Neutrophils (10^9/L): >13.5 | 0 | 0
  Lymphocytes (10^9/L): <0.8: number analyzed (Participants) | 98 | 113
  Lymphocytes (10^9/L): <0.8 | 13 | 15
  Lymphocytes (10^9/L): >12: number analyzed (Participants) | 98 | 113
  Lymphocytes (10^9/L): >12 | 1 | 0
  Monocytes (10^9/L): >2.5: number analyzed (Participants) | 98 | 113
  Monocytes (10^9/L): >2.5 | 0 | 0
  Eosinophils (10^9/L): >1.6: number analyzed (Participants) | 98 | 113
  Eosinophils (10^9/L): >1.6 | 1 | 0
  Basophils (10^9/L): >1.6: number analyzed (Participants) | 98 | 113
  Basophils (10^9/L): >1.6 | 0 | 0
  Hemoglobin (g/L): <=95 (F) or <=115 (M): number analyzed (Participants) | 98 | 113
  Hemoglobin (g/L): <=95 (F) or <=115 (M) | 0 | 2
  Hemoglobin (g/L): >=175 (F) or >=190 (M): number analyzed (Participants) | 98 | 113
  Hemoglobin (g/L): >=175 (F) or >=190 (M) | 0 | 0
  Hematocrit (%): <=32 (F) or <=37 (M): number analyzed (Participants) | 98 | 113
  Hematocrit (%): <=32 (F) or <=37 (M) | 2 | 5
  Hematocrit (%): >=54 (F) or >=60 (M): number analyzed (Participants) | 98 | 113
  Hematocrit (%): >=54 (F) or >=60 (M) | 0 | 0
  Red blood cells (10^12/L): <=3.5: number analyzed (Participants) | 98 | 113
  Red blood cells (10^12/L): <=3.5 | 0 | 0
  Red blood cells (10^12/L): >=6.4: number analyzed (Participants) | 98 | 113
  Red blood cells (10^12/L): >=6.4 | 0 | 0
  Platelets (10^9/L): <=75: number analyzed (Participants) | 98 | 113
  Platelets (10^9/L): <=75 | 0 | 0
  Platelets (10^9/L): >=700: number analyzed (Participants) | 98 | 113
  Platelets (10^9/L): >=700 | 0 | 0
  Sodium (mmol/L): <=126 | 0 | 0
  Sodium (mmol/L): >=156 | 0 | 0
  Potassium (mmol/L): <=3 | 0 | 1
  Potassium (mmol/L): >=6 | 0 | 0
  Chloride (mmol/L): <=90 | 0 | 0
  Chloride (mmol/L): >=118 | 0 | 0
  Bicarbonate (mmol/L): <=16 | 1 | 1
  Bicarbonate (mmol/L): >=35 | 0 | 0
  Calcium (mmol/L): <=2 | 0 | 1
  Calcium (mmol/L): >=3 | 0 | 0
  Phosphorus (mmol/L): <=0.5491 | 0 | 1
  Phosphorus (mmol/L): >=1.7119 | 0 | 0
  Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT): >=3xULN | 0 | 0
  Alanine aminotransferase (ALT)/serum glutamate pyruvate transaminase (SGPT): >=3xULN | 0 | 0
  Alkaline phosphatase: >=3xULN | 0 | 0
  Creatinine: >=1.5xULN | 0 | 0
  Total bilirubin: >=1.5xULN | 0 | 1
  Total protein (g/L): <=45 | 0 | 0
  Total protein (g/L): >=100 | 0 | 0
  Albumin (g/L): <=25 | 0 | 0
  Uric acid (umol)/L: >=501.5 (F) or >=619.5 (M) | 1 | 0
  Glucose (non-fasting) (mmol/L): <=2.2 | 0 | 0
  Glucose (non-fasting) (mmol/L): >=13.75 | 1 | 1

15. Secondary Outcome: Part 2: Number of Participants With Potentially Clinically Significant Electrocardiogram (ECG) Values
Description: The ECG result was classified as "normal", "abnormal", "abnormal, not adverse event", or "abnormal, adverse event". Shift to 'abnormal, not adverse event' included shift from normal or unknown to 'abnormal, not adverse event'. Shift to 'abnormal, adverse event' included shift from normal or unknown to 'abnormal, adverse event'.
Time Frame: Part 2: Baseline to Week 96
Population: Safety population included all participants who received at least 1 dose of study treatment. Participants were analyzed based on the actual treatment allocation. 'Number Analyzed' signifies number of participants analyzed at the specified timepoint for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo to BIIB033 750 mg | Part 2: BIIB033 750 mg
Number analyzed (Participants) | 100 | 113
Participants
  At Day 1: Normal | 83 | 89
  At Day 1: Abnormal, not Adverse Event | 10 | 16
  From Day 1 to Week 12: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 80 | 82
  From Day 1 to Week 12: Shift to Abnormal, not Adverse Event | 7 | 6
  From Day 1 to Week 12: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 80 | 82
  From Day 1 to Week 12: Shift to Abnormal, Adverse Event | 1 | 0
  From Day 1 to Week 24: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 79 | 88
  From Day 1 to Week 24: Shift to Abnormal, not Adverse Event | 4 | 8
  From Day 1 to Week 24: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 79 | 88
  From Day 1 to Week 24: Shift to Abnormal, Adverse Event | 0 | 0
  From Day 1 to Week 36: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 75 | 85
  From Day 1 to Week 36: Shift to Abnormal, not Adverse Event | 3 | 10
  From Day 1 to Week 36: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 75 | 85
  From Day 1 to Week 36: Shift to Abnormal, Adverse Event | 0 | 1
  From Day 1 to Week 48: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 71 | 79
  From Day 1 to Week 48: Shift to Abnormal, not Adverse Event | 2 | 7
  From Day 1 to Week 48: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 71 | 79
  From Day 1 to Week 48: Shift to Abnormal, Adverse Event | 0 | 1
  From Day 1 to Week 60: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 52 | 50
  From Day 1 to Week 60: Shift to Abnormal, not Adverse Event | 3 | 5
  From Day 1 to Week 60: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 52 | 50
  From Day 1 to Week 60: Shift to Abnormal, Adverse Event | 0 | 0
  From Day 1 to Week 72: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 23 | 23
  From Day 1 to Week 72: Shift to Abnormal, not Adverse Event | 1 | 2
  From Day 1 to Week 72: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 23 | 23
  From Day 1 to Week 72: Shift to Abnormal, Adverse Event | 0 | 0
  From Day 1 to Week 84: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 4 | 8
  From Day 1 to Week 84: Shift to Abnormal, not Adverse Event | 0 | 2
  From Day 1 to Week 84: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 4 | 8
  From Day 1 to Week 84: Shift to Abnormal, Adverse Event | 0 | 0
  From Day 1 to Week 96: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 2 | 0
  From Day 1 to Week 96: Shift to Abnormal, not Adverse Event | 0 |
  From Day 1 to Week 96: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 2 | 0
  From Day 1 to Week 96: Shift to Abnormal, Adverse Event | 0 |
  At Week 12: Normal | 80 | 81
  At Week 12: Abnormal, not Adverse Event | 9 | 16
  At Week 12: Abnormal, Adverse Event | 1 | 0
  From Week 12 to Week 24: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 79 | 87
  From Week 12 to Week 24: Shift to Abnormal, not Adverse Event | 4 | 7
  From Week 12 to Week 24: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 79 | 87
  From Week 12 to Week 24: Shift to Abnormal, Adverse Event | 0 | 0
  From Week 12 to Week 36: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 76 | 86
  From Week 12 to Week 36: Shift to Abnormal, not Adverse Event | 4 | 8
  From Week 12 to Week 36: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 76 | 86
  From Week 12 to Week 36: Shift to Abnormal, Adverse Event | 0 | 0
  From Week 12 to Week 48: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 73 | 81
  From Week 12 to Week 48: Shift to Abnormal, not Adverse Event | 3 | 6
  From Week 12 to Week 48: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 73 | 81
  From Week 12 to Week 48: Shift to Abnormal, Adverse Event | 0 | 2
  From Week 12 to Week 60: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 54 | 52
  From Week 12 to Week 60: Shift to Abnormal, not Adverse Event | 5 | 5
  From Week 12 to Week 60: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 54 | 52
  From Week 12 to Week 60: Shift to Abnormal, Adverse Event | 0 | 0
  From Week 12 to Week 72: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 26 | 24
  From Week 12 to Week 72: Shift to Abnormal, not Adverse Event | 2 | 1
  From Week 12 to Week 72: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 26 | 24
  From Week 12 to Week 72: Shift to Abnormal, Adverse Event | 0 | 0
  From Week 12 to Week 84: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 6 | 7
  From Week 12 to Week 84: Shift to Abnormal, not Adverse Event | 0 | 2
  From Week 12 to Week 84: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 6 | 7
  From Week 12 to Week 84: Shift to Abnormal, Adverse Event | 0 | 0
  From Week 12 to Week 96: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 2 | 0
  From Week 12 to Week 96: Shift to Abnormal, not Adverse Event | 0 |
  From Week 12 to Week 96: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 2 | 0
  From Week 12 to Week 96: Shift to Abnormal, Adverse Event | 0 |
  At Week 24: Normal | 83 | 83
  At Week 24: Abnormal, not Adverse Event | 6 | 20
  From Week 24 to Week 36: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 78 | 81
  From Week 24 to Week 36: Shift to Abnormal, not Adverse Event | 5 | 4
  From Week 24 to Week 36: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 78 | 81
  From Week 24 to Week 36: Shift to Abnormal, Adverse Event | 0 | 1
  From Week 24 to Week 48: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 74 | 77
  From Week 24 to Week 48: Shift to Abnormal, not Adverse Event | 1 | 5
  From Week 24 to Week 48: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 74 | 77
  From Week 24 to Week 48: Shift to Abnormal, Adverse Event | 0 | 1
  From Week 24 to Week 60: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 56 | 50
  From Week 24 to Week 60: Shift to Abnormal, not Adverse Event | 4 | 3
  From Week 24 to Week 60: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 56 | 50
  From Week 24 to Week 60: Shift to Abnormal, Adverse Event | 0 | 0
  From Week 24 to Week 72: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 27 | 22
  From Week 24 to Week 72: Shift to Abnormal, not Adverse Event | 2 | 1
  From Week 24 to Week 72: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 27 | 22
  From Week 24 to Week 72: Shift to Abnormal, Adverse Event | 0 | 0
  From Week 24 to Week 84: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 6 | 5
  From Week 24 to Week 84: Shift to Abnormal, not Adverse Event | 0 | 2
  From Week 24 to Week 84: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 6 | 5
  From Week 24 to Week 84: Shift to Abnormal, Adverse Event | 0 | 0
  From Week 24 to Week 96: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 3 | 0
  From Week 24 to Week 96: Shift to Abnormal, not Adverse Event | 0 |
  From Week 24 to Week 96: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 3 | 0
  From Week 24 to Week 96: Shift to Abnormal, Adverse Event | 0 |
  At Week 36: Normal | 77 | 80
  At Week 36: Abnormal, not Adverse Event | 7 | 20
  At Week 36: Abnormal, Adverse Event | 0 | 1
  From Week 36 to Week 48: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 75 | 75
  From Week 36 to Week 48: Shift to Abnormal, not Adverse Event | 3 | 3
  From Week 36 to Week 48: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 75 | 75
  From Week 36 to Week 48: Shift to Abnormal, Adverse Event | 0 | 2
  From Week 36 to Week 60: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 57 | 51
  From Week 36 to Week 60: Shift to Abnormal, not Adverse Event | 6 | 5
  From Week 36 to Week 60: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 57 | 51
  From Week 36 to Week 60: Shift to Abnormal, Adverse Event | 0 | 0
  From Week 36 to Week 72: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 26 | 24
  From Week 36 to Week 72: Shift to Abnormal, not Adverse Event | 2 | 1
  From Week 36 to Week 72: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 26 | 24
  From Week 36 to Week 72: Shift to Abnormal, Adverse Event | 0 | 0
  From Week 36 to Week 84: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 5 | 7
  From Week 36 to Week 84: Shift to Abnormal, not Adverse Event | 0 | 2
  From Week 36 to Week 84: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 5 | 7
  From Week 36 to Week 84: Shift to Abnormal, Adverse Event | 0 | 0
  From Week 36 to Week 96: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 3 | 0
  From Week 36 to Week 96: Shift to Abnormal, not Adverse Event | 0 |
  From Week 36 to Week 96: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 3 | 0
  From Week 36 to Week 96: Shift to Abnormal, Adverse Event | 0 |
  At Week 48: Normal | 74 | 76
  At Week 48: Abnormal, not Adverse Event | 4 | 15
  At Week 48: Abnormal, Adverse Event | 0 | 2
  From Week 48 to Week 60: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 56 | 52
  From Week 48 to Week 60: Shift to Abnormal, not Adverse Event | 4 | 4
  From Week 48 to Week 60: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 56 | 52
  From Week 48 to Week 60: Shift to Abnormal, Adverse Event | 0 | 0
  From Week 48 to Week 72: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 27 | 24
  From Week 48 to Week 72: Shift to Abnormal, not Adverse Event | 2 | 2
  From Week 48 to Week 72: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 27 | 24
  From Week 48 to Week 72: Shift to Abnormal, Adverse Event | 0 | 0
  From Week 48 to Week 84: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 6 | 8
  From Week 48 to Week 84: Shift to Abnormal, not Adverse Event | 0 | 1
  From Week 48 to Week 84: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 6 | 8
  From Week 48 to Week 84: Shift to Abnormal, Adverse Event | 0 | 0
  From Week 48 to Week 96: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 3 | 0
  From Week 48 to Week 96: Shift to Abnormal, not Adverse Event | 0 |
  From Week 48 to Week 96: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 3 | 0
  From Week 48 to Week 96: Shift to Abnormal, Adverse Event | 0 |
  At Week 60: Normal | 53 | 52
  At Week 60: Abnormal, not Adverse Event | 6 | 10
  From Week 60 to Week 72: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 26 | 24
  From Week 60 to Week 72: Shift to Abnormal, not Adverse Event | 1 | 2
  From Week 60 to Week 72: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 26 | 24
  From Week 60 to Week 72: Shift to Abnormal, Adverse Event | 0 | 0
  From Week 60 to Week 84: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 6 | 7
  From Week 60 to Week 84: Shift to Abnormal, not Adverse Event | 0 | 2
  From Week 60 to Week 84: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 6 | 7
  From Week 60 to Week 84: Shift to Abnormal, Adverse Event | 0 | 0
  From Week 60 to Week 96: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 2 | 0
  From Week 60 to Week 96: Shift to Abnormal, not Adverse Event | 0 |
  From Week 60 to Week 96: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 2 | 0
  From Week 60 to Week 96: Shift to Abnormal, Adverse Event | 0 |
  At Week 72: Normal | 26 | 24
  At Week 72: Abnormal, not Adverse Event | 2 | 4
  From Week 72 to Week 84: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 5 | 7
  From Week 72 to Week 84: Shift to Abnormal, not Adverse Event | 0 | 1
  From Week 72 to Week 84: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 5 | 7
  From Week 72 to Week 84: Shift to Abnormal, Adverse Event | 0 | 0
  From Week 72 to Week 96: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 2 | 0
  From Week 72 to Week 96: Shift to Abnormal, not Adverse Event | 0 |
  From Week 72 to Week 96: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 2 | 0
  From Week 72 to Week 96: Shift to Abnormal, Adverse Event | 0 |
  At Week 84: Normal | 7 | 7
  At Week 84: Abnormal, not Adverse Event | 0 | 3
  From Week 84 to Week 96: Shift to Abnormal, not Adverse Event: number analyzed (Participants) | 3 | 0
  From Week 84 to Week 96: Shift to Abnormal, not Adverse Event | 0 |
  From Week 84 to Week 96: Shift to Abnormal, Adverse Event: number analyzed (Participants) | 3 | 0
  From Week 84 to Week 96: Shift to Abnormal, Adverse Event | 0 |
  At Week 96: Normal | 3 | 0
  At Week 96: Abnormal, not Adverse Event | 0 | 1

16. Secondary Outcome: Part 2: Percentage of Participants With Potentially Clinically Significant Abnormal Vital Signs Values
Description: Vital sign measurements including temperature, pulse rate (supine), systolic blood pressure (BP) and diastolic (supine) BP were evaluated for safety. Criteria for abnormalities: Temperature: >38 degree celsius (◦C) or >=1 ◦C increase from baseline (BL); Pulse: [>100 beats per minute (bpm) or increase from BL of >30 bpm] or (<40 bpm or decrease from BL of >20 bpm); Systolic BP: [>160 millimeters of mercury (mmHg)/increase from BL of >40 mmHg] or (<90 mmHg/decrease from BL of >30 mmHg); Diastolic BP: (>100 mmHg/increase from BL of >30 mmHg) or (<45 mmHg/decrease from BL of >20 mmHg).
Time Frame: Part 2: Baseline to Week 96
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: Placebo to BIIB033 750 mg | Part 2: BIIB033 750 mg
Number analyzed (Participants) | 100 | 113
percentage of participants
  Temperature: >38 ◦C or >=1 ◦C Increase From BL | 4 | 5
  Pulse: (>100 bpm or increase from BL of >30 bpm) or (<40 bpm or decrease from BL of >20 bpm) | 22 | 25
  Pulse: >100 bpm or >30 bpm increase from BL | 11 | 15
  Pulse: <40 bpm or >20 bpm decrease from BL | 13 | 11
  Systolic BP: (>160 mmHg/increase from BL of >40 mmHg) or (<90 mmHg/decrease from BL of >30 mmHg) | 8 | 10
  Systolic BP: >160 mmHg or >40 mmHg increase from BL | 4 | 4
  Systolic BP: <90 mmHg or >30 mmHg decrease from BL | 4 | 8
  Diastolic BP: (>100 mmHg/increase from BL of >30 mmHg) or (<45 mmHg/decrease from BL of >20 mmHg) | 13 | 9
  Diastolic BP: >100 mmHg or >30 mmHg increase from BL | 3 | 4
  Diastolic BP: <45 mmHg or >20 mmHg decrease from BL | 11 | 5

17. Secondary Outcome: Part 2: Percentage of Participants With Potentially Clinically Significant Abnormal Weight Values
Description: Criteria for abnormality was defined as a >7% increase or decrease in weight at the specified time point.
Time Frame: Part 2: Baseline, Week 12, 24, 36, 48, 72 and 96
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: Placebo to BIIB033 750 mg | Part 2: BIIB033 750 mg
Number analyzed (Participants) | 100 | 113
percentage of participants
  At Baseline with Increase >7%: number analyzed (Participants) | 97 | 112
  At Baseline with Increase >7% | 27 | 15
  At Baseline with Decrease >7%: number analyzed (Participants) | 97 | 112
  At Baseline with Decrease >7% | 4 | 15
  At Week 12 with Increase >7%: number analyzed (Participants) | 89 | 101
  At Week 12 with Increase >7% | 4 | 3
  At Week 12 with Decrease >7%: number analyzed (Participants) | 89 | 101
  At Week 12 with Decrease >7% | 1 | 2
  At Week 24 with Increase >7%: number analyzed (Participants) | 92 | 104
  At Week 24 with Increase >7% | 10 | 10
  At Week 24 with Decrease >7%: number analyzed (Participants) | 92 | 104
  At Week 24 with Decrease >7% | 1 | 5
  At Week 36 with Increase >7%: number analyzed (Participants) | 87 | 103
  At Week 36 with Increase >7% | 18 | 5
  At Week 36 with Decrease >7%: number analyzed (Participants) | 87 | 103
  At Week 36 with Decrease >7% | 1 | 7
  At Week 48 with Increase >7%: number analyzed (Participants) | 79 | 96
  At Week 48 with Increase >7% | 20 | 8
  At Week 48 with Decrease >7%: number analyzed (Participants) | 79 | 96
  At Week 48 with Decrease >7% | 0 | 10
  At Week 72 with Increase >7%: number analyzed (Participants) | 59 | 66
  At Week 72 with Increase >7% | 19 | 15
  At Week 72 with Decrease >7%: number analyzed (Participants) | 59 | 66
  At Week 72 with Decrease >7% | 3 | 12
  At Week 96 with Increase >7%: number analyzed (Participants) | 27 | 31
  At Week 96 with Increase >7% | 30 | 13
  At Week 96 with Decrease >7%: number analyzed (Participants) | 27 | 31
  At Week 96 with Decrease >7% | 4 | 16

18. Secondary Outcome: Part 2: Number of Participants With Columbia Suicide Severity Rating Scale (C-SSRS) Score at Any Post-Baseline Visit
Description: C-SSRS systematically assess suicidal ideation and behavior rating scale. It rates an individual's degree of suicidal ideation on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent and behaviors". The scale identifies specific behaviors ranging from "preparatory acts or behavior" to "suicide" which may be indicative of an individual's intent to complete suicide.
Time Frame: Part 2: Baseline to Week 96
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo to BIIB033 750 mg | Part 2: BIIB033 750 mg
Number analyzed (Participants) | 100 | 113
Participants
  Suicidal Ideation: Wish to be Dead: number analyzed (Participants) | 98 | 113
  Suicidal Ideation: Wish to be Dead | 2 | 3
  Suicidal Ideation: Non-specific Active Suicidal Thoughts: number analyzed (Participants) | 98 | 113
  Suicidal Ideation: Non-specific Active Suicidal Thoughts | 0 | 1
  Suicidal Ideation: Active Suicidal Ideation with any Methods (not Plan) Without Intent to act: number analyzed (Participants) | 98 | 113
  Suicidal Ideation: Active Suicidal Ideation with any Methods (not Plan) Without Intent to act | 0 | 1
  Suicidal Ideation: Active Suicidal Ideation with Some Intent to act, Without Specific Plan: number analyzed (Participants) | 98 | 113
  Suicidal Ideation: Active Suicidal Ideation with Some Intent to act, Without Specific Plan | 0 | 1
  Suicidal Ideation: Active Suicidal Ideation with Specific Plan and Intent: number analyzed (Participants) | 98 | 113
  Suicidal Ideation: Active Suicidal Ideation with Specific Plan and Intent | 0 | 1
  Suicidal Behavior: Preparatory Acts or Behavior: number analyzed (Participants) | 98 | 113
  Suicidal Behavior: Preparatory Acts or Behavior | 0 | 1
  Suicidal Behavior: Aborted Attempt: number analyzed (Participants) | 98 | 113
  Suicidal Behavior: Aborted Attempt | 0 | 1
  Suicidal Behavior: Interrupted Attempt: number analyzed (Participants) | 98 | 113
  Suicidal Behavior: Interrupted Attempt | 0 | 1
  Suicidal Behavior: Actual Attempt: number analyzed (Participants) | 98 | 113
  Suicidal Behavior: Actual Attempt | 0 | 1
  Suicidal Behavior: Suicidal Behavior: number analyzed (Participants) | 98 | 113
  Suicidal Behavior: Suicidal Behavior | 0 | 1
  Suicidal Behavior: Suicide: number analyzed (Participants) | 97 | 112
  Suicidal Behavior: Suicide | 0 | 0
  Self-injurious Behavior Without Suicidal Intent: number analyzed (Participants) | 98 | 113
  Self-injurious Behavior Without Suicidal Intent | 0 | 0

ADVERSE EVENTS:
Time Frame: Part 1: From first dose through 12 weeks after administration of the last dose of study treatment (Up to Week 84); Part 2: From first dose through 12 weeks after administration of the last dose of study treatment (Up to Week 169)
Description: Safety population included all participants who received at least 1 dose of study treatment. Participants were analyzed based on the actual treatment allocation.
Arm/Group | Part 1: Placebo | Part 1: BIIB033 750 mg | Part 2: Placebo to BIIB033 750 mg | Part 2: BIIB033 750 mg
All-Cause Mortality (participants affected / at risk) | 0/131 | 1/132 | 0/100 | 0/113
Serious Adverse Events (participants affected / at risk) | 6/131 | 9/132 | 9/100 | 2/113
Other Adverse Events (participants affected / at risk) | 91/131 | 93/132 | 34/100 | 46/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo (N=131) | Part 1: BIIB033 750 mg (N=132) | Part 2: Placebo to BIIB033 750 mg (N=100) | Part 2: BIIB033 750 mg (N=113)
Congenital anomaly (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Coeliac artery compression syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Pelvic abscess (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Multiple sclerosis relapse (Nervous system disorders) | 1 | 0 | 0 | 0
Uhthoff's phenomenon (Nervous system disorders) | 1 | 0 | 0 | 0
Alcohol use disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Adenomyosis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Systemic infection (Infections and infestations) | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Chronic lymphocytic leukaemia stage 1 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Meningocele acquired (Nervous system disorders) | 0 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo (N=131) | Part 1: BIIB033 750 mg (N=132) | Part 2: Placebo to BIIB033 750 mg (N=100) | Part 2: BIIB033 750 mg (N=113)
Diarrhoea (Gastrointestinal disorders) | 11 | 6 | 3 | 6
Nausea (Gastrointestinal disorders) | 10 | 11 | 0 | 0
Vomiting (Gastrointestinal disorders) | 7 | 4 | 0 | 0
Fatigue (General disorders) | 14 | 14 | 0 | 0
Bronchitis (Infections and infestations) | 6 | 10 | 0 | 0
Nasopharyngitis (Infections and infestations) | 30 | 26 | 4 | 7
Sinusitis (Infections and infestations) | 5 | 9 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 20 | 31 | 5 | 9
Urinary tract infection (Infections and infestations) | 19 | 18 | 6 | 10
Fall (Injury, poisoning and procedural complications) | 12 | 17 | 4 | 8
Weight increased (Investigations) | 3 | 8 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 8 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 8 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 2 | 5 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 10 | 0 | 0
Dizziness (Nervous system disorders) | 9 | 5 | 0 | 0
Headache (Nervous system disorders) | 23 | 19 | 11 | 9
Multiple sclerosis relapse (Nervous system disorders) | 20 | 23 | 12 | 13
Paraesthesia (Nervous system disorders) | 8 | 7 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 9 | 0 | 0

LIMITATIONS AND CAVEATS:
The top-line results from the Part 1 did not meet the pre-specified primary endpoint nor the key secondary endpoints. The decision to discontinue study 215MS202 Part 2 was not based on safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for non-commercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/73/NCT03222973/Prot_002.pdf
  • Statistical Analysis Plan (2020-07-31): https://cdn.clinicaltrials.gov/large-docs/73/NCT03222973/SAP_003.pdf